CLINICAL TRIAL: NCT00833430
Title: Hedrocel Avascular Necrosis (AVN) Intervention Implant
Brief Title: Avascular Necrosis (AVN) Long-Term Follow-up
Status: Terminated | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: IC006-99
Record Dates: First submitted 2009-01-28; First posted 2009-02-02 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Avascular Necrosis; Femoral Head Collapse
Keywords: AVN; Femoral Head Collapse
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Long-term follow-up of IDE patients for publication

DETAILED DESCRIPTION:
This device (Hedrocel AVN Intervention Implant) was approved via 510(k) on April 15, 2005. One site was left open to follow patients to 5 year follow-up for publication of device survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Patient qualifies for core decompression based on physical exam
* No history of core decompression
* Patient is willing and able to provide written informed consent

Exclusion Criteria:

* Patient has been diagnosed as Stage 0, III, IV, V or VI using the Steinberg/UPenn staging system.
* Patient's BMI is >40
* Patient is mentally compromised
* Patient has neurological condition in ipsilateral or contralateral limb, which affect lower limb function
* The patient has had a proximal femoral osteotomy or internal fixation in the affected hip.
* The patient has undergone previous treatment for AVN
* Previous hip conditions
* Patient's bone stock is insufficient
* Patient has diagnosed systemic disease
* Patient is a pregnant female
* Patient is unable or unwilling to attend postop follow-up visits
* Patient has received investigational drug within the previous 6 months or an investigational device within the last 12 months
* Patient has an active or latent infection
* Patient has metal sensitivity
* Patient is a prisoner

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients enrolled at investigational sites who had Stage I or Stage II Osteonecrosis of the femoral head and who would qualify for core decompression based upon physical and radiographic exam and medical history.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2006-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety, Efficacy and longevity of device with patient as opposed to conventional total hip replacement | 5 Year Follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Emory Orthopedic Clinic, Atlanta, Georgia, United States